CLINICAL TRIAL: NCT00557609
Title: A Phase 2 Study of ARQ 197 in Patients With Microphthalmia Transcription Factor Associated Tumors
Brief Title: Phase 2 Study in Patients With MiT Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-204
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Renal Cell Carcinoma (RCC); Alveolar Soft Part Sarcoma (ASPS); Clear Cell Sarcoma (CCS)
Keywords: Microphthalmia transcription (MiT) factor associated tumors; Alveolar soft part sarcoma (ASPS); Clear cell sarcoma (CCS); Renal cell carcinoma (RCC)
MeSH Terms: conditions — Carcinoma, Renal Cell; Sarcoma, Alveolar Soft Part; Sarcoma, Clear Cell | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ARQ 197 — 360 mg administered twice daily until disease progression or other discontinuation criterion is met

SUMMARY:
This is a multi-center, single arm intended to evaluate the anti-tumor effect of ARQ 197 in patients with microphthalmia transcription factor associated (MiT) tumors. MiT tumors include clear cell sarcoma, alveolar soft parts sarcoma, and translocation associated renal cell carcinoma.

DETAILED DESCRIPTION:
This is a multi-center, single arm, two-stage phase 2 study of ARQ 197 in patients with microphthalmia transcription factor associated (MiT) tumors. ARQ 197 is a novel small molecule drug designed to block the activity of c-Met, which is thought to play multiple key roles in human cancer, including cancer cell growth, survival, angiogenesis, invasion and metastasis.

The microphthalmia transcription factor tumors (MiT tumors) are clear cell sarcoma (CCS), alveolar soft part sarcoma (ASPS), and translocation associated renal cell carcinoma (RCC). These soft tissue cancers are characterized by a common transcriptional mechanism that leads to inexorable spread and resistance to all known therapies. They tend to strike adolescents and young adults, and are invariably fatal if not resectable at diagnosis. Several academic laboratories have shown that genetic translocations in these tumors upregulate c-Met, and that such tumors are dependent upon this activity.

The study will enroll adolescent (age 13 or older) and adult patients with a histologically or cytologically confirmed MiT malignant disease. Eligible patients will receive ARQ 197 twice daily. Treatment will be continued until progression of disease, unacceptable toxicity, or another discontinuation criterion is met.

During the study, tumor evaluations will be performed at baseline, then in 8-week intervals.

To evaluate each patient's safety and the drug's toxicity, physical examinations, laboratory evaluations, vitals signs, and adverse event assessments will be performed throughout the study. Blood samples for PK analysis will be collected during first cycle of treatment from up to 10 patients aged 20 or younger. Archival tissue specimens and relevant laboratory results on patients' gene translocation/fusion status will be collected.

Tumor biopsies may also be collected (optional) with patient's consent. If patients agree tumor samples may be collected using core needle biopsy.

In addition, to explore biological responses of tumors to ARQ 197 treatment, FDG-PET scanning will be performed at three time points: within 14 days prior to the treatment, on Day 8 (± 2 days) of Cycle 1 and after two cycles of treatment coinciding with tumor measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed unresectable locally advanced or metastatic alveolar soft part sarcoma, clear cell sarcoma, or translocation associated renal cell carcinoma
2. ≥13 years old
3. Male or female patients of child-producing potential must agree to use double barrier contraception, oral contraceptives or avoidance of pregnancy measures during the study and for 30 days after the last ARQ 197 dose
4. Females of childbearing potential must have a negative serum pregnancy test

Exclusion Criteria:

1. Central nervous system metastasis unless it has been stable for ≥ 3 months after treatment and patient has no neural symptoms
2. Pregnant or lactating
3. Significant gastrointestinal disorder(s), in the opinion of a Investigator, could interfere with the absorption of ARQ 197 (e.g., Crohn's disease, ulcerative colitis, extensive gastric or small bowel resection)
4. Unable or unwilling to swallow ARQ 197 capsules twice daily
5. Known human immunodeficiency virus (HIV), Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
6. Bradycardia at baseline or known history of arrhythmia
7. Received ARQ 197 previously

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Determine the overall response rate (ORR) in patients treated with ARQ 197

SECONDARY OUTCOMES:
Evaluate progression-free survival (PFS) time in patients treated with ARQ 197
Evaluate 6-month and 1-year overall survival (OS) rates in patients treated with ARQ 197
Further characterize the safety of ARQ 197 in adolescent and young adult patients with MiT tumors

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - San Francisco, California
  - Santa Monica, California
  - Miami, Florida
  - Boston, Massachusetts
  - Cincinnati, Ohio
  - Dallas, Texas
  - Houston, Texas
- Toronto, Ontario, Canada
- London, United Kingdom

REFERENCES:
- [Derived] Wagner AJ, Goldberg JM, Dubois SG, Choy E, Rosen L, Pappo A, Geller J, Judson I, Hogg D, Senzer N, Davis IJ, Chai F, Waghorne C, Schwartz B, Demetri GD. Tivantinib (ARQ 197), a selective inhibitor of MET, in patients with microphthalmia transcription factor-associated tumors: results of a multicenter phase 2 trial. Cancer. 2012 Dec 1;118(23):5894-902. doi: 10.1002/cncr.27582. Epub 2012 May 17. PMID 22605650